CLINICAL TRIAL: NCT04076774
Title: A Functional Performance Study of The Wondaleaf Female Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Mags Beksinska (Other)
Responsible Party: Sponsor-Investigator, Prof Mags Beksinska, Deputy Executive Director, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MD20180502; 5020 (Registry Identifier: South African Clinical Trials Registry)
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: HIV Prevention; Pregnancy Prevention
Keywords: female condom; HIV and STI prevention; Condom acceptability; Wondaleaf; FC2

STUDY DESIGN:
Intervention Model Description: This research study will be a two-period, cross-over randomized controlled trial to compare the functional performance, safety and acceptability of two FC types (FC2 and Wondaleaf).
Who Masked: Outcomes Assessor
Masking Description: The two devices in the trial are distinctly different and so device specific training is required and so cannot be blinded. The statistician analysing the data will be blinded to female condom type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Wondaleaf female condom (Experimental): Participants will be provided with 5 Wondaleaf condoms first at enrolment and switched to 5 FC2 condoms at the first follow up visit
  Interventions: Device: Wondaleaf Female Condom; Device: FC2 Female Condom
- FC2 Female condom (Active Comparator): Participants will be provided with 5 FC2 condoms first at enrolment and switched to 5 Wondaleaf condoms at the first follow up visit
  Interventions: Device: Wondaleaf Female Condom; Device: FC2 Female Condom

INTERVENTIONS:
Device: Wondaleaf Female Condom — Wondaleaf: Wondaleaf is an ultra thin (of 0.02 mm) polyurethane female/male condom (16x8cm) that has folded extended adhesive shields (front 18x18cm, back 18x10cm), which at unfolding covers the entire external genitalia to prevent direct skin contact and exchange of body fluid between sexual partners during intercourse. Insertion of the condom body into the vagina is through use of a small medical grade cotton tissue packed inside the foil package. This is inserted into the end of the condom body and used to push the condom into the vagina. Each condom is individually packaged without prior lubrication. However, lubricant is expected to be used at donning the condom and during sexual intercourse. The lubricant will be supplied in separate packets together with the condom. Unlike latex, polyurethane condoms are unlikely to cause any allergic reaction and are much stronger than conventional latex condoms
Device: FC2 Female Condom — FC2: The FC2 is a second-generation female condom manufactured by the Female Health Company (Chicago, IL). The FC2 has US FDA approval and has been granted the CE Mark (Conformité Européenne) of the European Union. The FC2 is the only female condom that has been pre-qualified by the World Health Organisation. The device is similar in design to the FC1, but is made from a synthetic polymer (nitrile) film that is softer and more elastic than the polyurethane of the earlier device. The condom is designed as a loose-fitting pouch that lines the vagina. It has two flexible rings. The outer ring at the open end is rolled from the nitrile material. The outer ring remains outside the vagina and covers the external genitalia during intercourse. An internal polyurethane ring is removable and serves as the insertion mechanism and anchors the device within the vagina. FC2 measures 180mm in length and 80mm in lay-flat width. The device is pre-lubricated with dimethicone.

SUMMARY:
This research study will determine how well two female condoms perform when used during sex. One of these condoms (FC2) is already commercially available in South Africa. The other female condom, "Wondaleaf Condom" is a new female condom. Participants will use both condoms. The study aims to determine how well these condoms work comparatively. Study visits include a screening/enrolment visit and 2 follow up visits.

DETAILED DESCRIPTION:
This research study will determine how well two female condoms perform when used during sex. One of these condoms (FC2) is already commercially available in South Africa. The other female condom, "Wondaleaf Condom" is a new female condom. Participants will use both condoms. The study aims to determine how well these condoms work comparatively.

The Wondaleaf female condom is a new female condom (FC) design made of polyurethane with no external or internal rings. The body of the condom is fitted by an exterior adhesive shield which also displays the condom when removed from the condom packaging.

Purpose: To ascertain the functional performance of the Wondaleaf FC. This research study will be a two-period, cross-over randomized controlled trial to compare the functional performance, safety and acceptability of two FC types.

Study Design: The study will enrol 220 women, anticipating that 200 participants complete the study. The age range of these participants is from 18-45 years. Each participant will be asked to use five Wondaleaf FCs and five FC2 female condoms (available in the South African public sector).

Primary endpoints will be total clinical failure and total device failure for each condom type. Secondary endpoints will include rates of invagination, complete slippage, misdirection, and breakage.

Function, safety, and acceptability will be assessed at two follow-up visits approximately one month apart after enrollment. Participants will complete a Condom Log at home which gathers data on experience after use of each condom.

Female clients of the Commercial City Clinic will be told about the study. If a potential participant expresses interest in participating, the participant will be given the study information to read, which will describe the study requirements and the potential role in the study. If the participant agrees to take part in the research, the participant will be asked to provide written consent. The participant will be screened to ensure that the requirements for study participation are met.

Enrolled participants will be asked to use five FC2 and five Wondaleaf FCs. Participants will be asked to return to the clinic for follow-up after using each type of device. During the 1st follow-up visit, participants will be interviewed about the first assigned condom type and will receive the next condom packet within their second assigned (randomized) use sequence. In the second follow-up visit, participants will be interviewed about use of the condoms and will be discontinued from study participation. Data on device function, safety and acceptability for each condom type will be collected during follow-up visits.

At enrolment, baseline data will be gathered on participant demographics and past FC use via the baseline questionnaire. Using a pelvic model, the study staff will demonstrate female condom insertion and train the participants in the proper use of the first assigned female condom. Further, study staff will re- emphasize the instructions on how to complete the condom use log. Participants will be told that they do not have to use the FCs during consecutive acts of intercourse. The study staff will discuss with the participant an approximate timeframe for use of all 5 condoms and a suitable follow-up date will be scheduled. This date will be noted on an appointment slip. Participants will be encouraged to come back if condoms are finished before the due date and will be given the research study contact details to call for any appointment changes.

Follow-up visits: There will be two follow-up visits. During the first follow-up visit, study staff will review the information on the Condom Use Logs for completeness and accuracy. Further, the participants will be asked questions from a follow-up survey about the experiences using the FCs. Participants will be trained in the use of the second condom type, and given appropriate written condom use instructions. Staff will schedule the second follow-up visit, and participants will obtain the next condom packet in the assigned use sequence. At the end of the second follow-up visit the discontinuation form will be completed. Participation period for study participants is expected to last between 2-4 months.

The study will be registered on the South African clinical trials registry (SANCTR) and on clinicaltrials.gov.

The study will be monitored by an independent monitor contracted by the study investigator. The monitoring visit schedule includes an initiation visit, one interim visit and a close out visit. Risk based monitoring will be conducted for the study. The following study records will be reviewed:

* 100% of informed consent forms
* 100% of 100 enrolled participant files for source data verification
* 100% of serious adverse events and protocol deviations
* Investigator site file
* Study product No audits are planned for the study. The study has employed data staff to complete daily quality control of documents to ensure accuracy and completeness of data and electronic case report forms.

The site has Standard Operating Procedures in place to ensure consistency of site operations and study procedures. In addition, a source document guide and Manual of Procedures will be developed to ensure conformity.

Statistical Considerations:

The hypothesis for the primary endpoints, total clinical failure and total failure of a female condom and their components, is that the new condom WC2 is 'non-inferior' to FC2 with regard to the rate of events within a margin of 3.0%. That is, that the rate of events of each of the new condoms is not worse than that of the FC2 by more than 3.0%.

To demonstrate non-inferiority at a 5% significance level, the study will require the upper limit of the one-sided 95% confidence interval or equivalently the upper limit of the two-sided 90% confidence interval for the difference in the occurrence of events (New - FC2) to be below 3.0%.

It was calculated that the power to demonstrate non-inferiority obtained for different sample sizes, starting by the minimum of 200 couples completing the study recommended by ISO standards. It was assumed a total failure rate of 4% for the FC2 as reported from past research. It was assumed a correlation between uses of 0.15, as reported for male condoms. This assumption is more conservative than the maximum of 0.20 recommended by International Organization for Standardization (ISO) standards for female condoms.

For acceptability, scores ranging from 1 (lowest) to 5 (highest) to be compared across condom types using Friedman test, the proposed sample size will provide more than 99% power to detect a minimum difference of 1 in the scores of any two condom types, in a 5% significance level two-sided test. This calculation assumes a standard error of 1 and adjusts for multiple inferences using Bonferroni criterion, but ignores clustering (condoms within couples).

Data Analysis All analyses for primary and secondary endpoints will be performed according to the assigned condom use sequence among the subset of participants who provide relevant follow-up data on at least one condom of each type, no matter if they followed the assigned sequence. This will be the main analysis. An additional analysis will be performed with protocol compliers (i.e. participants who follow the assigned condom use sequence). All analyses for secondary endpoints will use a nominal 5% significance level.

A detailed analysis plan will be developed prior to the initiation of study enrollment. Any deviations to be made from this summary will be documented in the detailed analysis plan.

Condom Function The failure rates, or proportions of condom uses with clinical breakage, total breakage, slippage, misdirection, invagination, total clinical failure, and total FC failure will be summarized by condom type according to endpoint definitions. 95% confidence intervals for the proportion of each endpoint will be calculated using the exact method based on the binomial distribution.

Safety Data The proportion of participants with symptoms of genitourinary irritation during or immediately after any of the 5 separate uses and medical and serious adverse events, classified by relatedness to condom type, expectedness and severity will be reported.

Product Acceptability The key acceptability endpoints (listed below) will be summarized.

* comfort in use;
* ease of insertion and removal;
* like or dislike of product attributes and adequacy and feel of lubrication.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 45 years (inclusive);
2. Be literate (able to read a newspaper or letter easily);
3. Be sexually active (defined as having at least two vaginal coital acts per week and not being abstinent in the month prior to enrolment);
4. Be in an exclusive (monogamous) sexual relationship with her spouse or partner while participating in this research study;
5. Have been in a sexual relationship with this partner for at least 6 months;
6. Not be a sex worker;
7. Not be pregnant (as determined by pregnancy testing) or planning a pregnancy during the time of the research study;
8. Be without observable evidence of Sexually Transmitted Infections (STI) as determined through syndromic diagnosis and vaginal examination;
9. Be using hormonal or other non-barrier contraception (e.g. Oral Contraception (OCs), injectable, implant, Intra Uterine Device (IUD), or have had a tubal sterilization);
10. Not be menopausal (defined as 12 months without menstruation);
11. Not have had a hysterectomy;
12. Not have known sensitivities or allergies to latex, polyurethane, vaginal/sexual lubricants or the lubricants used on condoms;
13. Willing to give informed consent;
14. Willing to complete the FC coital use logs;
15. Willing to use the study condoms as directed;
16. Willing to adhere to the follow-up schedule and all study procedures;
17. Willing to provide research study staff with an address, phone number or other locator information while participating in the study; and,
18. Willing to participate in the study for the duration of 10 condom uses (approximately 2-4 months.
19. Willing to have fingerprint scan to check for co-enrolment in other research projects

Exclusion Criteria:

* None specified

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be female as female condoms inserted vaginally are being evaluated
Enrollment: 220 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Clinical breakage | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Clinical breakage is defined as breakage during sexual intercourse or during withdrawal of the female condom from the vagina. Clinical breakage is breakage with potential adverse clinical consequences. The clinical breakage rate is calculated by dividing the number of female condoms reported to have broken during sexual intercourse or during withdrawal by the number of female condoms used during sexual intercourse.
Total breakage | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Total breakage is defined as the sum of all female condom breakages at any time before, during or after sexual intercourse. It includes both clinical breakages and non-clinical breakages. The total breakage rate is calculated by dividing the total number of female condoms that broke by the number of female condom packages opened
Slippage | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Slippage is defined as an instance when a female condom slips completely out of the vagina during sexual intercourse. The slippage rate is calculated by dividing the number of female condoms that slipped by the number of female condoms used during sexual intercourse.
Misdirection | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Invagination is defined as an instance when the external retention feature of the female condom is partially or fully pushed into the vagina during sexual intercourse. The invagination rate is calculated by dividing the number of events of invagination by the number of female condoms used during sexual intercourse.
Invagination | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Invagination is defined as an instance when the external retention feature of the female condom is partially or fully pushed into the vagina during sexual intercourse. The invagination rate is calculated by dividing the number of events of invagination by the number of female condoms used during sexual intercourse.
Total clinical failure | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Total clinical failure is defined as the sum of female condoms that clinically break or slip, or are associated with misdirection, invagination or any additional failure modes(s) identified in the risk assessment which results in the reduction of the female condom protective function. The total clinical failure rate is calculated by dividing the number of female condoms with a clinical failure by the number of female condoms used during sexual intercourse.
Total female condom failure | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Total female condom failure is defined as a female condom for which a non-clinical breakage, clinical breakage or slippage occurs, or is associated with misdirection, invagination or any additional failure modes(s) identified in the risk assessment. The female condom failure rate is calculated by dividing the number of female condoms that fail by the number of female condom packages opened.

SECONDARY OUTCOMES:
Safety (Adverse Events) | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Proportion of participants with symptoms of and proportion of Wondaleaf condom uses with reports of genitourinary irritation during or immediately after any of the 5 separate uses will be calculated. Medical and serious adverse events will be classified by relatedness, expectedness and severity.
Acceptability | Number of condoms allocated in each arm is 5. Duration of time these condoms will be used depends on the coital frequency of the couple. Therefore the duration of time in each arm is dependent on time take to use all 5 condoms. (approximately 3-6 weeks)
  Frequency of key acceptability endpoints will be calculated and include: comfort in use; ease of insertion and removal; like or dislike of product attributes; and adequacy and feel of lubrication

CONTACTS AND LOCATIONS:
Overall Officials: Mags E Beksinska, PhD, Principal Investigator — Maternal, Adolescent and Child Health Research Unit
Locations (1):
- MatCH Research Unit [Maternal, Adolescent and Child Health Research Unit], Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trussell J, Sturgen K, Strickler J, Dominik R. Comparative contraceptive efficacy of the female condom and other barrier methods. Fam Plann Perspect. 1994 Mar-Apr;26(2):66-72. PMID 8033980
- [Background] Soper DE, Shoupe D, Shangold GA, Shangold MM, Gutmann J, Mercer L. Prevention of vaginal trichomoniasis by compliant use of the female condom. Sex Transm Dis. 1993 May-Jun;20(3):137-9. doi: 10.1097/00007435-199305000-00003. PMID 8511706
- [Background] Fontanet AL, Saba J, Chandelying V, Sakondhavat C, Bhiraleus P, Rugpao S, Chongsomchai C, Kiriwat O, Tovanabutra S, Dally L, Lange JM, Rojanapithayakorn W. Protection against sexually transmitted diseases by granting sex workers in Thailand the choice of using the male or female condom: results from a randomized controlled trial. AIDS. 1998 Oct 1;12(14):1851-9. doi: 10.1097/00002030-199814000-00017. PMID 9792386
- [Background] French PP, Latka M, Gollub EL, Rogers C, Hoover DR, Stein ZA. Use-effectiveness of the female versus male condom in preventing sexually transmitted disease in women. Sex Transm Dis. 2003 May;30(5):433-9. doi: 10.1097/00007435-200305000-00010. PMID 12916135
- [Background] Hoke TH, Feldblum PJ, Van Damme K, Nasution MD, Grey TW, Wong EL, Ralimamonjy L, Raharimalala L, Rasamindrakotroka A. Temporal trends in sexually transmitted infection prevalence and condom use following introduction of the female condom to Madagascar sex workers. Int J STD AIDS. 2007 Jul;18(7):461-6. doi: 10.1258/095646207781147175. PMID 17623503
- [Background] PATH and United Nations Population Fund (UNFPA). Female condom: a powerful tool for protection. Seattle: UNFPA, PATH; 2006. Available at: http://www.unfpa.org/upload/lib_pub_file/617_filename_female_condom.pdf.
- [Background] World Health Organization (WHO), United States Agency for International Development, Johns Hopkins Bloomberg School of Public Health. Family Planning, A Global Handbook for Providers. Baltimore, MD: Information & Knowledge for Optimal Health (INFO) Project; 2008.
- [Background] Beksinska M, Smit J, Joanis C, Usher-Patel M, Potter W. Female condom technology: new products and regulatory issues. Contraception. 2011 Apr;83(4):316-21. doi: 10.1016/j.contraception.2010.07.022. Epub 2010 Sep 15. PMID 21397088
- [Background] Ting RS, Wong EL, Tnay JK. A pilot study on the functional performance and acceptability of an innovative female condom (Wondaleaf(R)) in Malaysia. Open Access J Contracept. 2018 Jan 24;9:11-20. doi: 10.2147/OAJC.S152505. eCollection 2018. PMID 29440937
- [Background] Beksinska M, Joanis C, Manning J, Smit J, Callahan M, Deperthes B, Usher-Patel M. Standardized definitions of failure modes for female condoms. Contraception. 2007 Apr;75(4):251-5. doi: 10.1016/j.contraception.2006.10.003. Epub 2007 Feb 7. PMID 17362701
- [Background] Gallo MF, Grimes DA, Schulz KF. Non-latex versus latex male condoms for contraception. Cochrane Database Syst Rev. 2003;(2):CD003550. doi: 10.1002/14651858.CD003550. PMID 12804475
- [Background] Williams, E., Experimental Designs Balanced for the Estimation of Residual Effects of Treatments. Australian Journal of Chemistry, 1949. 2(2): p. 149-168.
- [Background] STATA User's Guide. College Station, Texas, USA: StataCorp, LP.
- [Background] Beksinska ME, Piaggio G, Smit JA, Wu J, Zhang Y, Pienaar J, Greener R, Zhou Y, Joanis C. Performance and safety of the second-generation female condom (FC2) versus the Woman's, the VA worn-of-women, and the Cupid female condoms: a randomised controlled non-inferiority crossover trial. Lancet Glob Health. 2013 Sep;1(3):e146-52. doi: 10.1016/S2214-109X(13)70054-8. Epub 2013 Aug 23. PMID 25104263
- [Background] Joanis C, Beksinska M, Hart C, Tweedy K, Linda J, Smit J. Three new female condoms: which do South-African women prefer? Contraception. 2011 Mar;83(3):248-54. doi: 10.1016/j.contraception.2010.08.002. Epub 2010 Sep 17. PMID 21310287
- [Background] Taylor D. Issues in the design, analysis and interpretation of condom functionality studies. Contraception. 2009 Sep;80(3):237-44. doi: 10.1016/j.contraception.2009.03.004. Epub 2009 Apr 23. PMID 19698815
- [Background] ISO 29943-2:2017 Condoms -- Guidance on clinical studies -- Part 2: Female condoms, clinical function studies based on self-reports.
- [Derived] Beksinska M, Mphili N, Smit J. Functional performance of the Wondaleaf condom: A crossover, noninferiority, randomized clinical trial. Int J STD AIDS. 2023 Feb;34(2):114-121. doi: 10.1177/09564624221139899. Epub 2022 Nov 25. PMID 36426764